CLINICAL TRIAL: NCT02481765
Title: Phase I Trial of the Feasibility and Dose Tolerability of High Definition Transcranial Direct Current Stimulation in Healthy Adults and Children With Down Syndrome
Brief Title: Feasibility and Dose Tolerability of HD-tDCS in Healthy Adults and Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014-0262; A535100 (Other: UW, Madison); SMPH/NEUROLOGY/NEUROLOGY (Other: UW, Madison)
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: HD-tDCS (High definition transcranial direct current stimulation)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Direct current Stimulation (Experimental): High definition transcranial direct current stimulation (HD-tDCS)
  Interventions: Device: High definition transcranial direct current stimulation

INTERVENTIONS:
Device: High definition transcranial direct current stimulation
  Other Names: HD-tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a method which enables noninvasive electrical stimulation of the cortex via electrodes placed on the subject's skull. High definition tDCS (HD-tDCS) allows for precise generation of electrical fields over selected cortical areas using multiple electrodes. The purpose of this pilot trial is to study feasibility, tolerability, and safety of HD-tDCS administered daily for a total of 20 sessions in healthy adults and 5-10 year old children with Down syndrome.

PRIMARY OBJECTIVES Part I: To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in healthy adult subjects; Part II: After review of the safety data for Part I is completed and reviewed by the Data Safety Monitoring Committee and IRB, Part II will be initiated. To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in adult subjects with Down Syndrome.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a method which enables noninvasive electrical stimulation of the cortex via electrodes placed on the subject's skull. tDCS has been shown to improve motor learning, visuomotor coordination, probabilistic classification, boost memory in humans and was found to be well tolerated in children with early onset schizophrenia, continuous spike-wave in sleep (CSWS), refractory epilepsy and dystonia. The method has been approved for investigational purposes by the FDA. High definition tDCS (HD-tDCS) allows for precise generation of electrical fields over selected cortical areas using multiple electrodes. Positioning of the stimulating electrodes is determined with the help of MR brain images and appropriate modeling. The purpose of this pilot trial is to study feasibility, tolerability, and safety of HD-tDCS administered daily for a total of 20 sessions.

PRIMARY OBJECTIVES Part I: To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in healthy adult subjects; Part I will be defined to be positive if 5 healthy adults are accrued within the study period (12 months) and at least 4 of 5 participants have successful completion. Tolerability will be measured as the proportion of subjects able to complete 20 sessions on the assigned treatment within 6 weeks.

Part II: After review of the safety data for Part I is completed and reviewed by the Data Safety Monitoring Committee and IRB, Part II will be initiated. To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in pediatric subjects with Down Syndrome; Part II will be defined to be positive if 5 children with Down Syndrome are accrued within the study period (24 months) and at least 4 of 5 participants have successful completion. Tolerability will be measured as the proportion of subjects able to complete 20 sessions on the assigned treatment within 6 weeks.

SECONDARY OBJECTIVES Part I: - Collect pilot data on safety of HD-tDCS in healthy adults, where safety is defined by incidents of adverse events. Safety outcomes will include vital signs, physical/neurologic exam findings, weight, electrocardiograms and electroencephalograms.

- Collect pilot data on feasibility of efficacy endpoints. These will include assessment of impact of HD-tDCS, administered up to 5 days per week for a total of 20 sessions, on EEG amplitudes and coherences in the lower (<8Hz) and higher (>9Hz) frequency ranges and coherences in the lower (<8Hz) and gamma (30-80 Hz) frequency ranges in healthy adults.

Part II: - Collect pilot data on safety of HD-tDCS in children (5-10 years) with Down Syndrome, where safety is defined by incidents of adverse events. Procedures to monitor subject safety include vital sign measurements, physical/neurologic examinations, electrocardiograms and electroencephalograms. Clinically significant changes in the safety measures will be documented as adverse events.

Collect pilot data on feasibility of efficacy endpoints. These will include assessment of impact of HD-tDCS, administered up to 5 days per week for a total of 20 sessions, on EEG amplitudes and coherences in the lower (<8Hz) and higher (>9Hz) frequency ranges and coherences in the lower (<8Hz) and gamma (30-80 Hz) frequency ranges in children with Down Syndrome.

ELIGIBILITY:
PART I

Inclusion Criteria:

* Adult aged > 18 years and ≤ 45 years
* Healthy Adult subjects have the ability to consent for themselves.

No previous or current medical history of epilepsy, neurologic, heart, endocrinologic, renal, chronic infectious, metabolic, psychiatric disease or cancer

* Normal physical examination
* Normal neurologic examination
* Normal EKG
* Normal EEG
* IQ above 80. We will only include individuals with college education to assure that IQ requirements are met.

Exclusion Criteria:

* Previous or current medical history of epilepsy, neurologic, heart, endocrinologic, renal, chronic infectious, metabolic, psychiatric disease or cancer
* Healthy adult subjects will be excluded from the study if the subject is not suitable for study participation due to other reasons, at the discretion of the PI.

PART II

Inclusion criteria

* Adult aged > 18 years and ≤ 45 years
* Genetically confirmed Trisomy 21

Exclusion criteria

* Cardiac, hematologic, oncologic comorbidities that require intensive medical treatment. Intensive medical treatment means that the subject is undergoing chemotherapy for a hematologic/oncologic condition, is carrying a pacemaker or has been diagnosed with a cardiac anomaly which causes cardiac insufficiency not compensated with medications.
* Active epilepsy, history of epilepsy, history of seizures or with epileptiform discharges on screening baseline EEG.
* Anticipated inability of the subject to comply with the rigors of the protocol as outlined in the consent form.
* Behavioral problems of sufficient magnitude to preclude participation in the study. These include anxiety, obsessive compulsive behaviors, attention problems, agitation, oppositional behavior. These behavioral problems will be assessed during the first visit and the PI will make decision to exclude subjects which she considers will not be able to complete the study.
* The subject is legally blind (vision acuity <20/200 not correctable with lenses, as determined be a certified optometrist or an ophthalmologist).
* The subject is severely hearing impaired (Hearing level >71 dB, as measured with a standard audiometer at frequencies between 8 and 20 kHz).
* The subject is not suitable for study participation due to other reasons, at the discretion of the PI.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Feasibility and tolerability of HD-tDCS in healthy adult subjects | One year
  To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in healthy adult subjects; Part I will be defined to be positive if 5 healthy adults are accrued within the study period (12 months) and 4 of 5 participants (80%) have successful completion.
Feasibility and tolerability of HD-tDCS in adults with Down syndrome | Two years
  To assess feasibility and tolerability of HD-tDCS, administered up to 5 days per week for a total of 20 sessions in adult subjects with Down Syndrome; Part II will be defined to be positive if 5 adults with Down Syndrome are accrued within the study period (12 months) and at least 4 of 5 participants (80%) have successful completion.

SECONDARY OUTCOMES:
Collect pilot data on safety of HD-tDCS in healthy adults | One year
  Collect pilot data on safety of HD-tDCS in healthy adults, where safety is defined by incidence of adverse events.
Collect pilot data on feasibility of efficacy endpoints | One year
  - Collect pilot data on feasibility of efficacy endpoints. These will include assessment of impact of HD-tDCS, administered up to 5 days per week for a total of 20 sessions, on EEG amplitudes and coherences in healthy adults
Collect pilot data on safety of HD-tDCS in adults with Down Syndrome | Two years
  Collect pilot data on safety of HD-tDCS in adults with Down Syndrome, where safety is defined by incidence of adverse events.
Collect pilot data on feasibility of efficacy endpoints. | Two years
  - Collect pilot data on feasibility of efficacy endpoints. These will include assessment of impact of HD-tDCS, administered up to 5 days per week for a total of 20 sessions, on EEG amplitudes and coherences.

CONTACTS AND LOCATIONS:
Overall Officials: Hrissanthi Ikonomidou, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Neurology, University of Wisconsin Madison, Madison, Wisconsin, United States

REFERENCES:
- [Result] Turski CA, Kessler-Jones A, Chow C, Hermann B, Hsu D, Jones J, Seeger SK, Chappell R, Boly M, Ikonomidou C. Extended Multiple-Field High-Definition transcranial direct current stimulation (HD-tDCS) is well tolerated and safe in healthy adults. Restor Neurol Neurosci. 2017;35(6):631-642. doi: 10.3233/RNN-170757. PMID 29172010